CLINICAL TRIAL: NCT05519345
Title: Conditioning Brain Responses for Modulating Corticospinal Excitability After ACL Reconstruction
Brief Title: Operant Conditioning After ACL Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Riann Palmieri-Smith, Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00166442
Record Dates: First submitted 2022-08-17; First posted 2022-08-29 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Anterior Cruciate Ligament Injuries
Keywords: ACL; Quadriceps
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Operant Conditioning (Experimental): Motor evoked responses will be elicited along with operant conditioning training for about 2 weeks
  Interventions: Behavioral: Operant Conditioning
- Control (Experimental): Motor evoked responses will be elicited without operant conditioning training for about 2 weeks
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Operant Conditioning — Active encouragement and feedback to increase motor evoked response during stimulation.
  Arms: Operant Conditioning
Behavioral: Control — Absence of active encouragement and feedback to increase motor evoked response when stimulated.
  Arms: Control

SUMMARY:
The purpose of this study is to examine if the changes in corticospinal function that accompany ACL reconstruction can be improved through a form of mental coaching and encouragement, known as operant conditioning.

DETAILED DESCRIPTION:
It is theorized reduced corticospinal excitability contributes to quadriceps dysfunction after knee injury and joint disease. Current rehabilitation does not directly target the alterations in corticospinal excitability, which may limit recovery. Operant conditioning is an emerging approach capable of increasing corticospinal excitability by directly targeting the corticospinal pathways. However, it remains to be determined whether operant conditioning of the corticospinal pathway may improve corticospinal function after knee trauma. Therefore, this study will evaluate the ability of operant up-conditioning of the corticospinal pathway to improve corticospinal function after ACL reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* aged 14-45 years
* suffered an acute, complete ACL rupture
* have undergone ACL reconstructive surgery
* willingness to participate in testing and follow-up as outlined in the protocol

Exclusion Criteria:

* have suffered a previous ACL injury on the contralateral leg
* have undergone previous major surgery to the contralateral knee
* have a history of recent significant knee injury (other than ACL) or lower-extremity fracture
* have a history of uncontrolled diabetes or hypertension
* be pregnant or plan to become pregnant
* have metal implants in the head
* have electronic devices in their ear or heart (e.g., cochlear implants or cardiac pacemakers)
* have unexplained recurrent headaches
* have a recent history of seizure
* have a history of repeated fainting spells

Ages: 14 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2022-12-28 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2023-10-10 (Actual)

PRIMARY OUTCOMES:
Changes in corticospinal excitability | Baseline (before the start of the intervention) and post-intervention (approximately 2 weeks after baseline)
  Corticospinal excitability will be measured using transcranial magnetic stimulation at baseline and post-intervention and will be compared between groups.

OTHER OUTCOMES:
Changes in quadriceps strength | Baseline (before the start of the intervention) and post-intervention (approximately 2 weeks after baseline)
  Isometric quadriceps strength will be measured using an isokinetic dynamometer. Quadriceps strength will be measured prior to the intervention and immediately following the intervention.
Changes in quadriceps voluntary activation | Baseline (before the start of the intervention) and post-intervention (approximately 2 weeks after baseline)
  Voluntary activation will be measured using an electrical superimposition technique. Voluntary activation will be measured prior to the intervention and immediately following the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided